CLINICAL TRIAL: NCT05660590
Title: The Effect of Complex Decongestive Physiotherapy Applied With Different Compression Pressures on Skin and Subcutaneous Tissue Thickness in Individuals With Breast Cancer-related Lymphedema: a Double-blinded Randomized Comparison Trial
Brief Title: Effect of Different Bandage Interface Pressures on Breast Cancer Related Lymphedema
Acronym: BCRL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Elif Duygu, Research assistant, Abant Izzet Baysal University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BAIBU-FTR-ED-001
Record Dates: First submitted 2022-12-02; First posted 2022-12-21 (Actual); Last update posted 2022-12-29 (Actual); Status verified 2022-12

CONDITIONS: Lymphedema of Upper Limb; Breast Cancer Lymphedema; Edema Arm
Keywords: compelex decongestive physiotherapy; bandage interface pressure; compression therapy
MeSH Terms: conditions — Breast Cancer Lymphedema

STUDY DESIGN:
Intervention Model Description: Randomised comparison trial
Who Masked: Participant, Outcomes Assessor
Masking Description: radiologist who assessed soft tissue thickness assessment is masked and the patients did't know which group they belong to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low bandage pressure (Active Comparator): Compression bandages applied with low pressure (20-30 mmHg)
  Interventions: Other: complex decongestive physiotherapy with low pressure compression bandage
- high bandage pressure (Active Comparator): Compression bandages applied with low pressure (45-55 mmHg)
  Interventions: Other: complex decongestive physiotherapy with high pressure compression bandage

INTERVENTIONS:
Other: complex decongestive physiotherapy with low pressure compression bandage — both group received complex decongestive physiotherapy consist of manual lymph dranaige, skin care, exercise and compression bandage. Every component except compression bandage applied exacly the same to both group. Compression bandage applied with low bandage interface pressure (20-30 mmHg)
  Other Names: Low bandage interface pressure
  Arms: Low bandage pressure
Other: complex decongestive physiotherapy with high pressure compression bandage — complex decongestive physiotherapy consist of manual lymph dranaige, skin care, exercise and compression bandage. Every component except compression bandage applied exacly the same to both group. Compression bandage applied with high bandage interface pressure (45-55 mmHg)
  Other Names: High bandage interface pressure
  Arms: high bandage pressure

SUMMARY:
The goal of this randomised comparison study is to compare different bandage interface pressures in individuals with breast cancer related lymphedema

The main questions it aims to answer are:

* Is high or low bandage pressure effective in reducing edema and soft tissue thickness?
* do bandages applied with high or low bandage pressure comprimise sleep, comfort or subjective benefit from treatment?

Participants will recieve complex decongestive physiotherapy. Bandage will apply high or low pressure. Effects of high and low bandage interface pressures will compare

DETAILED DESCRIPTION:
The aim of this study was to evaluate the effect of compression bandage applied with different pressures on skin and subcutaneous thickness in individuals with breast cancer-related lymphedema.

individuals with stage 2 unilateral lymphedema participated in the study. Skin and subcutaneous thicknesses, extremity volumes, sleep quality, treatment benefit, comfort during treatment were evaluated respectively by ultrasound from 6 reference points as dorsum of hand, wrist volar, forearm dorsum, forearm volar, arm dorsum, arm volar, volumetric measurement, Pittsburgh Sleep Quality Index, Patient Benefit Index-Lymphedema, and visual analog scale. Complex decongestive physiotherapy was applied to individuals randomly divided into two groups: low (20-30 mmHg) and high bandage pressure (45-55 mmHg). Individuals were evaluated before treatment, at 1st, 10th session, end of treatment, and at 3 months follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Stage 2 unilateral BCRL involving whole extremity according to ISL
* To be volunteer.

Exclusion Criteria:

* Acute deep vein thrombosis
* Acute soft tissue infection
* Peripheral artery disease in upper extremity
* Systemic diseases with peripheral edema (kidney, hearth insufficiency etc.),
* Allergy to materials used for treatment
* Mental diseases effect cooperation
* Sensory loss in the effected limb
* Open wound in the effected limb.

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2022-04-22 (Actual); Study Completion 2022-05-18 (Actual)

PRIMARY OUTCOMES:
change from baseline skin and subcutanetous thickness with 4 weeks treatment and follow up | baseline, 1.day, 2 weeks, 4 weeks, 3 months (follow-up)
  Evaluation of skin and subcutaneous tissue thickness and US evaluations were made by a radiologist using a 6-15 MHz linear probe with a LOGIQ US system. Skin and subcutaneous thickness were recorded as milimeter.
change from baseline residual volume with 4 weeks treatment and follow up | baseline, 1.day, 2 weeks, 4 weeks, 3 months (follow-up)
  Limb volume was determined by the overflowing water method. The volumetric vessel was filled with tap water up to the overflow point of the vessel. Subjects were asked to lean forward while standing and slowly dip their arms into the water until the bar at the base of the volumetric cup snapped between the 2nd and 3rd fingers. During immersion, he was asked to avoid movements that could increase the transport of water. The overflowing water was first taken into a container. Then, the overflow water was calculated by transferring it to the measuring cups. The amount of overflowing water was recorded in ml. Measurements were made bilaterally.

SECONDARY OUTCOMES:
sleep quality | baseline, 4 weeks, 3 months (follow-up)
  Sleep quality was assessed with the Pittsburgh Sleep Quality Index (PSQI). The scale that determines sleep quality consists of 18 questions and evaluates sleep quality in the last four weeks. PSQI has 7 components, and each component is evaluated between 0-3 points. The total score ranges from 0-21 (206). A total score higher than 5 indicates poor sleep quality (28). The sub-dimensions of PSQI are subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbance, use of sleeping pills, and daytime dysfunction
Comfort | baseline, 4 weeks, 3 months (follow-up)
  Patient comfort was evaluated with Visual Analogue Scale at the end of the treatment. It was explained to the individual that 0 point of a 10 cm line represents minimum comfort and 10 point represents maximum comfort. The individual was asked to mark the level of comfort he perceived during the treatment. The point marked by the individual was measured with a ruler and recorded in cm.
Subjective benefit from treatment | 4 weeks
  The benefit from the treatment was evaluated with the Patient Benefit Index-Lymphedema. It consists of two five-point Likert-type questionnaires containing the same 23 questions, the Patient Needs Questionnaire, and the Patient Benefit Questionnaire. Scores of Index are between 0-4. "0" means no benefit from treatment. "4" means maximum benefit from treatment.
  score

CONTACTS AND LOCATIONS:
Overall Officials: elif duygu yıldız, Dr, Principal Investigator — Abant Izzet Baysal University
Locations (1):
- Abany Izzet Baysal University, Bolu, Center, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Duygu-Yildiz E, Bakar Y, Hizal M. The effect of complex decongestive physiotherapy applied with different compression pressures on skin and subcutaneous tissue thickness in individuals with breast cancer-related lymphedema: a double-blinded randomized comparison trial. Support Care Cancer. 2023 Jun 7;31(7):383. doi: 10.1007/s00520-023-07843-y. PMID 37285046